CLINICAL TRIAL: NCT06293391
Title: The Impact of Patient Position Changes on Advanced Hemodynamic Indices in Laparoscopic and Open Major Abdominal Cancer Surgeries
Brief Title: The Effect of Patient Position Changes on Advanced Cardiac Indices in Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2022-11/2097
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Abdominal Cancer; Blood Pressure; Cardiac Indices
MeSH Terms: interventions — Supine Position; Head-Down Tilt

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ODM measurements of patients undergoing open surgery in supine and trendelenburg position: After intubation, serial ODM measurements were performed in the supine and trendelenburg position of the patient and CO: Cardiac output, FTc: Flow time corrected, PV: Peak velocity, SD: Stroke distance values were recorded.
  Interventions: Procedure: cardiac indices in supine and trendelenburg position
- ODM measurements of patients undergoing laparoscopic surgery in supine and trendelenburg position: After intubation, serial ODM measurements were performed in the supine and trendelenburg position of the patient and CO: Cardiac output, FTc: Flow time corrected, PV: Peak velocity, SD: Stroke distance values were recorded.
  Interventions: Procedure: cardiac indices in supine and trendelenburg position

INTERVENTIONS:
Procedure: cardiac indices in supine and trendelenburg position — Cardiac indices in supine and trendelenburg position in patients undergoing open or laparoscopic major cancer surgery

SUMMARY:
Esophageal Doppler Monitoring (Deltex CardioQ Esophageal Doppler Monitor, ODM) is used to manage patients' fluid therapy by non-invasively measuring continuous cardiac output with an esophageal probe. The aim of this study was to compare the effects of patient position changes on cardiac indices and vital signs in patients who underwent major abdominal cancer surgery with laparoscopic and open surgery using ODM.

DETAILED DESCRIPTION:
Patients who underwent major abdominal cancer surgery using ODM in the operating room of our hospital between November 2021 and November 2022 were identified from the Anesthesiology Clinic records and examined according to whether they were operated with open or closed (laparoscopic) methods. Demographic data, vital signs, amount of bleeding, type and amount of fluid administered, and the results of cardiac index measurements performed with the ODM device in the supine and trendelenburg positions (45 degrees) were analyzed. Parameters recorded with the ODM device; CO: Cardiac output, FTc: Flow time corrected, PV: Peak velocity, SD: Stroke distance.

ELIGIBILITY:
Inclusion Criteria:

* Elective operation
* ASA 1-4

Exclusion Criteria:

* Heart failure
* Valvular heart disease,
* Patients with symptomatic rhythm disturbances
* ODM placement contraindicated (coagulopathy, oesophageal varices, known aortic aneurysm)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients included in the study were intubated after standard anaesthesia induction with fentanyl 2 mcg/kg, propofol 2 mg/kg and rocuronium 0.6 mg/kg, and ODM was used for case follow-up. All patients were followed with standard 6% desflurane anaesthetic gas and intravenous infusion of remifentanil, a short-acting opioid, after intubation. Mean arterial pressure was kept in the range of 65-80 mmHg in all patients, tidal volume was adjusted as 6-8 ml/kg, peep (positive end expiratory pressure) as 0-6 cm H2O and respiratory frequency as 10-15 /min for normocapnia. After intubation, intraoperative ODM measurements and intraoperative ODM measurements were retrospectively scanned and recorded in the supine and 45-degree angle trendelenburg position.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Stroke Volume | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Flow time corrected | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Peak Velocity | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Stroke Distance | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Mean arterial pressure | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.
Pulse | Immediately after induction of anaesthesia and at any stable time during the case
  Measurement of cardiac output with the oesophageal doppler device immediately after induction of anaesthesia and in the middle of the case in both supine and trendelenburg position of the patient to see whether there is a significant difference in positional change.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal SAHIN, M.D, Principal Investigator — Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Locations (1):
- Dr.Abdurrahman Yurtaslan Ankara Oncology Train and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Heinink TP, Read DJ, Mitchell WK, Bhalla A, Lund JN, Phillips BE, Williams JP. Oesophageal Doppler guided optimization of cardiac output does not increase visceral microvascular blood flow in healthy volunteers. Clin Physiol Funct Imaging. 2018 Mar;38(2):213-219. doi: 10.1111/cpf.12401. Epub 2017 Feb 6. PMID 28168868
- [Result] Yonis H, Bitker L, Aublanc M, Perinel Ragey S, Riad Z, Lissonde F, Louf-Durier A, Debord S, Gobert F, Tapponnier R, Guerin C, Richard JC. Change in cardiac output during Trendelenburg maneuver is a reliable predictor of fluid responsiveness in patients with acute respiratory distress syndrome in the prone position under protective ventilation. Crit Care. 2017 Dec 5;21(1):295. doi: 10.1186/s13054-017-1881-0. PMID 29208025
- [Result] Haas S, Haese A, Goetz AE, Kubitz JC. Haemodynamics and cardiac function during robotic-assisted laparoscopic prostatectomy in steep Trendelenburg position. Int J Med Robot. 2011 Dec;7(4):408-13. doi: 10.1002/rcs.410. Epub 2011 Aug 3. PMID 21815239
- [Result] Conway DH, Hussain OA, Gall I. A comparison of noninvasive bioreactance with oesophageal Doppler estimation of stroke volume during open abdominal surgery: an observational study. Eur J Anaesthesiol. 2013 Aug;30(8):501-8. doi: 10.1097/EJA.0b013e3283603250. PMID 23549128
- [Result] Kaye AD, Vadivelu N, Ahuja N, Mitra S, Silasi D, Urman RD. Anesthetic considerations in robotic-assisted gynecologic surgery. Ochsner J. 2013 Winter;13(4):517-24. PMID 24358000
- [Result] Huang L, Critchley LA. An assessment of two Doppler-based monitors to track cardiac output changes in anaesthetised patients undergoing major surgery. Anaesth Intensive Care. 2014 Sep;42(5):631-9. doi: 10.1177/0310057X1404200514. PMID 25233178
- [Derived] Argun G, Sahin MK. The impact of patient position changes on advanced hemodynamic indices in laparoscopic and open major abdominal cancer surgeries: retrospective study. BMC Surg. 2025 Aug 6;25(1):341. doi: 10.1186/s12893-025-03064-8. PMID 40770328